CLINICAL TRIAL: NCT06469801
Title: Low-Field Bedside MRI for Detection of Acute Brain Injury in Pediatric Extracorporeal Membrane Oxygenation
Brief Title: ECMO ABI Detection With Hyperfine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jessica S. Wallisch, Pediatric Intensivist, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003208
Record Dates: First submitted 2024-06-12; First posted 2024-06-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Acute Brain Injury; Extracorporeal Membrane Oxygenation Complication; Hypoxia-Ischemia, Brain; Stroke, Acute
Keywords: Pediatric
MeSH Terms: conditions — Brain Injuries; Hypoxia-Ischemia, Brain; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Portable MRI Arm (Experimental): All subjects enrolled will be assigned to Arm 1
  Interventions: Device: Hyperfine

INTERVENTIONS:
Device: Hyperfine — Enrolled subjects will undergo a Hyperfine MRI exam, which is a portable, low-field MRI, at various timepoints during their clinical course on ECMO. Patients will undergo imaging within 36 hours of ECMO initiation/cannulation. Patients that remain on ECMO will have repeat imaging at 72-120 hours of ECMO therapy and again weekly for the duration of their ECMO course. Patients will also undergo a portable MRI within 24 hours of clinical head imaging, if applicable.

SUMMARY:
The primary objective is to characterize the prevalence and type of ABI following cannulation for pediatric patients who require ECMO support. The secondary objective is to describe the time course and rates of ABI using ultralow-field bedside MRI relative to both duration of ECMO support and clinical imaging obtained in routine care of pediatric ECMO patients.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is frequently used to treat refractory cardiovascular and/or respiratory failure. As the support modality has evolved, survival has significantly improved, yet there are high rates of acute brain injury (ABI) in this population due to disease, patient, and treatment factors. This results in significant morbidity and mortality. Specifically, thromboembolic, hypoxic-ischemic, and hemorrhagic complications occur during ECMO support, but the investigators are limited in the monitoring and diagnosis of ABI while on ECMO as currently available imaging modalities (i.e. ultrasound [US], computed tomography [CT]) have low sensitivity for early hypoxic, cerebrovascular, and ischemic brain injuries. The sensitivity of these modalities increases only when it is too late to effectively intervene. Standard magnetic resonance imaging (MRI) is the gold standard to diagnose stroke and ischemic brain injury but is incompatible with ECMO devices. Swoop (Hyperfine, Guilford, CT) is an FDA cleared ultralow-field portable MRI system that can be used at the bedside and has been studied in critically ill adults with various types of ABI. This novel bedside MRI has been safely operated in clinical environments with equipment that is typically not MRI compatible. A few adult and pediatric ECMO patients have undergone bedside brain MRIs showing feasibility. Yet, what remains unknown is the true prevalence and timing of hypoxic, cerebrovascular, and ischemic brain injuries in pediatric ECMO.

ELIGIBILITY:
Inclusion Criteria

* Participants that will be or are admitted to the Pediatric Intensive Care Unit, Cardiac Intensive Care Unit, or the Neonatal Intensive Care Unit
* Ages 0-17 years
* Participants that are at high risk for undergoing ECMO or are currently undergoing venovenous or venoarterial ECMO

  • High risk participants include, but are not limited to:
* Undergoing cardiac surgery
* Congenital heart disease
* Congenital diaphragmatic hernia
* Refractory hypoxemic and/or hypercarbic respiratory failure
* Vasoactive-refractory shock

Exclusion Criteria

* Pregnancy
* Active implants such as:

  * Pacemaker
  * Implanted defibrillator
  * Implanted insulin pump
  * Deep brain stimulator
  * Vagus nerve stimulator
  * Cochlear implant
  * Programmable shunt
* MRI incompatible surgical hardware (e.g., staples, screws, etc.)
* Metal-containing tattoos or permanent make-up on head or neck
* Suspected metal in eye, e.g.,
* Former or current welders, metal workers, or individuals with a metal injury
* Metal shrapnel
* Passive implants are considered MRI-conditional

Ages: 0 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the prevalence and type of ABI following cannulation for pediatric patients who require ECMO support. | Duration of ECMO treatment period, an average of <2 weeks
  Perform bedside MRI in pediatric ECMO patients treated in pediatric, cardiac, and neonatal intensive care units (ICUs) within 36 hours of cannulation. Determine rates of ABI (hypoxic, ischemic, cerebrovascular, and hemorrhagic injury along with assessment of cerebral edema and midline shift) in the pre- and peri-cannulation time periods. Correlate these imaging findings to rates of clinical neurological events (seizures, pupillary changes, focal neurological examination).

SECONDARY OUTCOMES:
Describe the time course and rates of ABI using ultralow-field bedside MRI relative to both duration of ECMO support and clinical imaging obtained in routine care of pediatric ECMO patients. | Duration of ECMO treatment period, an average of <2 weeks
  Obtain bedside MRI in pediatric ECMO patients treated in pediatric, cardiac or neonatal ICUs at 72-120 hours post-cannulation and weekly until decannulation. Quantify and compare rates of ABI between bedside MRI and CT or US as read by blinded neuroradiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Wallisch, MD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No